CLINICAL TRIAL: NCT05917717
Title: Cardiac Arrest Bundle of Care Trial
Acronym: CABARET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: University of Southampton (Other); South Central Ambulance service (Unknown); Hampshire and Isle of Wight air Ambulance (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CABARET
Record Dates: First submitted 2023-05-25; First posted 2023-06-26 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Cardiopulmonary Resuscitation; Cardiac Arrest; Out of Hospital Cardiac Arrest
Keywords: Cardiac Arrest; Mechanical CPR; Cardiopulmonary Resuscitation; Impedance threshold device; Active compression decompression CPR; Head up cardiopulmonary resuscitation (HUP-CPR)
MeSH Terms: conditions — Heart Arrest; Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Intervention Model Description: Pilot study - randomised controlled trial
Who Masked: Outcomes Assessor
Masking Description: The study team will not be blinded to which patients receive which arm of the trial and will be aware of what each service is delivering in each phase of the study. The research team carrying out the flow up will be blinded to the arm of the trial that the participant was in when they are collecting outcome and follow up data.
  It is impossible to blind the care providers.
  Participants will be blinded to which arm of the trial they were in (should they regain capacity).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (usual care) (No Intervention): Usual care for a cardiac arrest patient with no deviation.
- Intervention 'bundle of care' (Experimental): The clinical team will follow a specific sequence of actions using three devices (Elegard, Lucas-3, and ITD-16), in addition to standard CPR. Firstly, they will place the ITD onto the i-gel) or ETT, followed by the Elegard device and the LUCAS-3. The team will also place a cerebral saturation monitor on (Near-Infrared Spectroscopy (NIRS)) (if they have access to one). After 2 minutes of CPR via the LUCAS-3 with the ResQPOD-16 (ITD), the Elegard device will be turned on and activated to gradually elevate the head approximately 22cm from the ground to the back of the occiput. If necessary, the clinical team may choose to intubate the trachea at this point. Resuscitation will continue for at least 30 minutes or until ROSC is achieved. If ROSC is achieved, standard post ROSC guidelines will be followed.
  Interventions: Procedure: Neuroprotective 'bundle of care'

INTERVENTIONS:
Procedure: Neuroprotective 'bundle of care' — This includes the 3 devices:
  * Head up cardiopulmonary resuscitation (HUP-CPR)
  * Active compression decompression CPR
  * Impedance threshold device (ITD)
  Arms: Intervention 'bundle of care'

SUMMARY:
An out-of-hospital cardiac arrest is a sudden event where the heart stops beating and a person becomes unresponsive. During this event, vital organs in the body receive no blood flow, causing them to shut down. Without intervention to restart the heart, a person effectively dies. In the UK, around 60,000 people experience cardiac arrests each year, with most occurring at home. Despite prompt emergency service response, survival rates are typically low.

There is technology available that has the potential to improve survival rates for out-of-hospital cardiac arrests. The intervention involves three devices used together: head-up position CPR (Elegard), active compression-decompression mechanical CPR (Lucas-3), and the Impedance Threshold device (Resqpod-16). When combined, these devices can enhance blood flow during resuscitation, potentially leading to improved initial resuscitation rates and higher rates of survival with normal brain function after a cardiac arrest.

A pilot study is planned to test the feasibility of using these devices. The results will inform the design of a larger study to determine if this technology can indeed improve survival rates in out-of-hospital cardiac arrests.

DETAILED DESCRIPTION:
Out of hospital cardiac arrest (OOHCA) is the sudden cessation of effective cardiovascular circulation in the pre hospital setting. This is sadly a common occurrence within the UK with approximately 60,000 OOHCAs per year. In 30,000 of these, resuscitation is attempted by the ambulance service. Survival remains poor (2-12%) within the UK and even the best performing regions still lag someway behind exemplar global systems (Seattle 21%, Norway 25%). There are a plethora of reasons for variation in outcome, not limited to the availability of community defibrillators, the education and ability of bystanders to provide effective CPR, the response times of the emergency medical personnel, the training of emergency services personnel and their individual exposure to cardiac arrest, the availability of primary percutaneous coronary intervention, and even the availability of extracorporeal resuscitation.

Despite poor outcomes from OOHCA for decades, there exists promising data from animal and cadaver studies that new technological devices could improve the currently poor blood flow generated by chest compressions during CPR, particularly cerebral blood flow. The current standard of care for patients with an OOHCA includes manual CPR delivered at a rate of 100-120 compressions per minute with a depth of 5 cm (maximum 6 cm). In turn, periodic inflation of the lungs using positive pressure ventilation to maintain oxygenation is mandated during CPR. Animal data have shown that blood flow to the heart and brain using this method is approximately 15-30% of normal. Conventional CPR is therefore unphysiological by definition, with intracerebral pressures being too high in the compression phase and intrathoracic pressure being too high in the release phase for adequate blood flow to the brain and heart respectively. Mechanisms and tools to improve this have been available for some time but using them synergistically to achieve improved cerebral and coronary blood flow is a relatively recent advance.

It is now possible to mimic a more physiologically normal situation by combining 3 pieces of technology. These may lead to better organ perfusion during CPR and therefore better rates of survival. The 3 devices in question do this in different complementary ways, in turn;

1. Head up position- gradated elevation of the head after CPR has been initiated, improves cerebral blood flow during CPR. This has been studied predominantly in porcine models. HUP-CPR enhances venous return, and reduces intracranial pressure during the decompression phase of CPR. This results in improved cerebral perfusion pressure and improves cerebral blood flow.
2. Active compression/decompression CPR uses a device with a suction cup placed on the thorax that via active decompression generates a negative intrathoracic pressure on each upward stroke, meaning that venous return to the heart improves during each cycle of CPR, allowing more blood to then be pumped to the brain on the next compressive cycle.
3. Combined with an impedance threshold device which works by limiting air entry into the lungs during chest recoil between chest compressions thereby enhancing the lower intrathoracic pressure achieved by active decompression, as described above.

The first retrospective study examining the combination of active compression decompression CPR with an ITD and HUP-CPR in humans was published in 2022, concluding that rapid initiation of bundle of care-CPR was associated with a higher likelihood of survival to hospital discharge after OHCA when compared with conventional CPR. 9. The first prospective human study using this triple bundle approach is currently ongoing in France.

The 3 devices described above are all CE marked meaning that this trial is not a trial of an experimental device and therefore does not need to be reported to the MHRA for their regulatory approvals.

Justification for undertaking the trial

Survival from OOHCA in the UK remains extremely poor (2-12%). The fact that this has not changed over many decades is of concern. Additionally, the global health disparity that exists in survival from OOCHA between different healthcare systems is stark.

The published animal data has created a plausible biological signal that improvements with cerebral blood flow are indeed possible using a bundle approach to neuroprotective CPR. The practicalities of performing this in human subjects in cardiac arrest is already being done in certain emergency medical systems globally. One study has published retrospective data with a signal to suggest that improved outcomes are possible using this approach. As far as the investigators are aware, no randomised control trial is currently being undertaken to test this hypothesis.

The proposed treatment bundle holds the potential to change this, the investigators are of the opinion that this should be tested scientifically within the remit of a clinical trial and this is the first necessary stage of that process. The individual components have shown promise in animal studies but this has not been borne out in the human trials that have followed. The synergistic and complementary effect of the 3 devices that make up the bundle of care in this study have the potential to change outcomes.

In parts of the USA (Seattle and Phoenix Fire departments) this bundle of care has been brought in due to the marked improvements in survival that have been seen. The investigators are of the opinion that an adequately powered randomised trial is essential to confirm these possible benefits.

Research statement

Out-of-hospital cardiac arrest (OOHCA) is a common event with poor long-term survival rates, often resulting in poor neurological outcomes. While there are several interventions that may improve survival and neurological outcomes, single interventions alone have not consistently demonstrated significant improvements in outcomes. The combination of head up cardiopulmonary resuscitation (CPR), active compression decompression CPR, and the use of an impedance threshold device has not yet been tested in a pragmatic randomised controlled trial. Therefore, the objective of this study is to assess the feasibility of conducting a randomized trial comparing usual care with a "bundle of care" approach incorporating the above interventions to improve patient outcomes after OOHCA.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (>18 year of age) who have suffered a cardiac arrest
2. Body habitus is compatible with the bundle devices.
3. Witnessed event
4. Time of collapse was known with reasonable certainty to have been to be within 20 minutes.

Exclusion Criteria:

1. Visibly pregnant women
2. Prisoners
3. Traumatic cardiac arrest
4. Drowning
5. Hanging
6. DNACPR
7. Have been in witnessed cardiac arrest for an estimated time of 21 minutes or more

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-05-24 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
The feasibility of initiating the 'bundle of care' (ability to recruit to the intervention, ability to place the 3 devices in the intervention group and use them as per the protocol. | Through study completion an average of up to 1 year
  The feasibility of initiating the 'bundle of care' (ability to recruit to the intervention) and to adequately perform the randomisation and crossover of each arm within each participating service, evidenced by the number of eligible patients and the number recruited.
Feasibility of delivering a single education package on how to use the 'bundle of care'. | 30 days
  The feasibility of delivering an education package to teach the procedure for the bundle of care intervention and the success of said education package, evidenced by the number of staff trained and the incidence of non-compliance. The package will contain classroom teaching and video resources.

SECONDARY OUTCOMES:
First recorded cardiac rhythm of the participants in the trial | 30 Minutes
  To record the initial cardiac arrest rhythm, asystole, pulseless electrical activity, ventricular fibrillation or ventricular tachycardia.
Signs of life during CPR to include a pulse, an attempt to breathe or to move | 30 minutes
  Signs of life during CPR- Presence of agonal respirations and other signs of life (pupillary response, movement during CPR)
Maximum end tidal carbon dioxide (CO2) during CPR before ROSC. | 30 minutes
Return of spontaneous circulation (ROSC). | 60-120 minutes
  To mark the time of ROSC is it is achieved.
Is the participant alive at hospital at the point of handover in the emergency department (i.e. sustained ROSC) or are they dead. | 60-120 minutes
  Is the patient alive or dead, this is a binary outcome measure
To evaluate any differences between intubation and supraglottic airway use with regard to mortality. | 30 days
To evaluate any differences between intubation and supraglottic airway use with regard to modified Rankin score. | 30 days
  The Modified Rankin score is a score from 0-5 with a higher score indicating a worse neurological outcome after cardiac arrest. The values are as follows.
  0 The patient has no residual symptoms.
  1. The patient has no significant disability; able to carry out all pre-stroke activities.
  2. The patient has slight disability; unable to carry out all pre-stroke activities but able to look after self without daily help.
  3. The patient has moderate disability; requiring some external help but able to walk without the assistance of another individual.
  4. The patient has moderately severe disability; unable to walk or attend to bodily functions without assistance of another individual.
  5. The patient has severe disability; bedridden, incontinent, requires continuous care.
Survival to discharge or 30-day survival (whichever is sooner). | 30 days
Survival with a favourable neurological outcome at hospital discharge (or 30 days) using The modified Rankin Scale (mRS) | 30 days
  The Modified Rankin score is a score from 0-5 with a higher score indicating a worse neurological outcome after cardiac arrest. The values are as follows.
  0 The patient has no residual symptoms.
  1. The patient has no significant disability; able to carry out all pre-stroke activities.
  2. The patient has slight disability; unable to carry out all pre-stroke activities but able to look after self without daily help.
  3. The patient has moderate disability; requiring some external help but able to walk without the assistance of another individual.
  4. The patient has moderately severe disability; unable to walk or attend to bodily functions without assistance of another individual.
  5. The patient has severe disability; bedridden, incontinent, requires continuous care.
To complete a service user questionnaire on the delivery of the intervention. | 30 days
  To evaluate the opinions of the paramedics and doctors recruiting to the trial regarding the use of the equipment in the intervention group and any barriers to recruitment.

CONTACTS AND LOCATIONS:
Overall Officials: James Plumb, PhD, Principal Investigator — University Hospital Southampton NHS Foundation Trust
Locations (1):
- University Hospital Southampton NHS Foundation trust, Southampton, England, United Kingdom

IPD SHARING:
Plan to Share IPD: No
We will use this data to inform a definitive trial in this area

REFERENCES:
- [Background] Hawkes C, Booth S, Ji C, Brace-McDonnell SJ, Whittington A, Mapstone J, Cooke MW, Deakin CD, Gale CP, Fothergill R, Nolan JP, Rees N, Soar J, Siriwardena AN, Brown TP, Perkins GD; OHCAO collaborators. Epidemiology and outcomes from out-of-hospital cardiac arrests in England. Resuscitation. 2017 Jan;110:133-140. doi: 10.1016/j.resuscitation.2016.10.030. Epub 2016 Nov 17. PMID 27865775
- [Background] Berdowski J, Berg RA, Tijssen JG, Koster RW. Global incidences of out-of-hospital cardiac arrest and survival rates: Systematic review of 67 prospective studies. Resuscitation. 2010 Nov;81(11):1479-87. doi: 10.1016/j.resuscitation.2010.08.006. Epub 2010 Sep 9. PMID 20828914
- [Background] Perkins GD, Cooke MW. Variability in cardiac arrest survival: the NHS Ambulance Service Quality Indicators. Emerg Med J. 2012 Jan;29(1):3-5. doi: 10.1136/emermed-2011-200758. Epub 2011 Nov 1. No abstract available. PMID 22045608
- [Background] Lindner TW, Soreide E, Nilsen OB, Torunn MW, Lossius HM. Good outcome in every fourth resuscitation attempt is achievable--an Utstein template report from the Stavanger region. Resuscitation. 2011 Dec;82(12):1508-13. doi: 10.1016/j.resuscitation.2011.06.016. Epub 2011 Jun 24. PMID 21752524
- [Background] Moore JC, Salverda B, Rojas-Salvador C, Lick M, Debaty G, G Lurie K. Controlled sequential elevation of the head and thorax combined with active compression decompression cardiopulmonary resuscitation and an impedance threshold device improves neurological survival in a porcine model of cardiac arrest. Resuscitation. 2021 Jan;158:220-227. doi: 10.1016/j.resuscitation.2020.09.030. Epub 2020 Oct 4. PMID 33027619
- [Background] Moore JC, Segal N, Lick MC, Dodd KW, Salverda BJ, Hinke MB, Robinson AE, Debaty G, Lurie KG. Head and thorax elevation during active compression decompression cardiopulmonary resuscitation with an impedance threshold device improves cerebral perfusion in a swine model of prolonged cardiac arrest. Resuscitation. 2017 Dec;121:195-200. doi: 10.1016/j.resuscitation.2017.07.033. Epub 2017 Aug 5. PMID 28827197
- [Background] Kim DW, Choi JK, Won SH, Yun YJ, Jo YH, Park SM, Lee DK, Jang DH. A new variant position of head-up CPR may be associated with improvement in the measurements of cranial near-infrared spectroscopy suggestive of an increase in cerebral blood flow in non-traumatic out-of-hospital cardiac arrest patients: A prospective interventional pilot study. Resuscitation. 2022 Jun;175:159-166. doi: 10.1016/j.resuscitation.2022.03.032. Epub 2022 Apr 5. PMID 35395338
- [Background] Moore JC, Pepe PE, Scheppke KA, Lick C, Duval S, Holley J, Salverda B, Jacobs M, Nystrom P, Quinn R, Adams PJ, Hutchison M, Mason C, Martinez E, Mason S, Clift A, Antevy PM, Coyle C, Grizzard E, Garay S, Crowe RP, Lurie KG, Debaty GP, Labarere J. Head and thorax elevation during cardiopulmonary resuscitation using circulatory adjuncts is associated with improved survival. Resuscitation. 2022 Oct;179:9-17. doi: 10.1016/j.resuscitation.2022.07.039. Epub 2022 Aug 4. PMID 35933057
- [Background] Perkins GD, Handley AJ, Koster RW, Castren M, Smyth MA, Olasveengen T, Monsieurs KG, Raffay V, Grasner JT, Wenzel V, Ristagno G, Soar J; Adult basic life support and automated external defibrillation section Collaborators. European Resuscitation Council Guidelines for Resuscitation 2015: Section 2. Adult basic life support and automated external defibrillation. Resuscitation. 2015 Oct;95:81-99. doi: 10.1016/j.resuscitation.2015.07.015. Epub 2015 Oct 15. No abstract available. PMID 26477420
- [Background] Aufderheide TP, Nichol G, Rea TD, Brown SP, Leroux BG, Pepe PE, Kudenchuk PJ, Christenson J, Daya MR, Dorian P, Callaway CW, Idris AH, Andrusiek D, Stephens SW, Hostler D, Davis DP, Dunford JV, Pirrallo RG, Stiell IG, Clement CM, Craig A, Van Ottingham L, Schmidt TA, Wang HE, Weisfeldt ML, Ornato JP, Sopko G; Resuscitation Outcomes Consortium (ROC) Investigators. A trial of an impedance threshold device in out-of-hospital cardiac arrest. N Engl J Med. 2011 Sep 1;365(9):798-806. doi: 10.1056/NEJMoa1010821. PMID 21879897
- [Background] Wang CH, Tsai MS, Chang WT, Huang CH, Ma MH, Chen WJ, Fang CC, Chen SC, Lee CC. Active compression-decompression resuscitation and impedance threshold device for out-of-hospital cardiac arrest: a systematic review and metaanalysis of randomized controlled trials. Crit Care Med. 2015 Apr;43(4):889-96. doi: 10.1097/CCM.0000000000000820. PMID 25517475
- See also: Clinical trial - GRAVITY — https://clinicaltrials.gov/ct2/show/NCT03996616
- See also: King County 2013 Annual Report — http://www.google.com/search?q=D+F%2C+J+F.+Emergency+Medical+Services+Division+Of.%3B+2013.&rlz=1C5CHFA_enGB745GB745&oq=D+F%2C+J+F.+Emergency+Medical+Services+Division+Of.%3B+2013.&aqs=chrome..69i57j0i546j69i64.1166j0j4&sourceid=chrome&ie=UTF-8